CLINICAL TRIAL: NCT06767384
Title: Diagnostic Accuracy of x Ray Kub in Diagnosing Renal Calculi Keeping CT Scan as Gold Standard
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHS/Batch-Spring23/034
Record Dates: First submitted 2024-12-18; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Renal Calculi
MeSH Terms: conditions — Kidney Calculi | interventions — X-Rays

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: X-ray — To determine diagnostic accuracy of x-ray KUB in diagnostic renal and ureter calculi keeping CT scan KUB as a gold standard.

SUMMARY:
In clinical practice both Xray and CT Scan KUB are reliable,however, Ctscan is superior to X ray KUB in detecting renal and ureteric calculi,the reson being stone that are missed by xray KUB are usually small and sould pass spontenously while other are usually with improper bowel preparation

ELIGIBILITY:
Inclusion Criteria:

* Female who will be advised X ray KUB and CT scan KUB for suspected renal & uretrric calculi(flank pain )for <24 hours .
* Age 18-49 years (because this is common age group for renal &ureteric calculi).

Exclusion criteria:

* Female patients with pregnancy.
* Morbidly obese patients (Men>129 kg women>113kg)
* Patients with history of any abdominal trauma

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Aim is to check the Diagnostic Accuracy of x Ray Kub in Diagnosing Renal Calculi Keeping CT Scan as Gold Standard
Sampling Method: Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
multidetector computed tomography | 12 Months
  multidetector computed tomography scan Kidney UreterBladder

CONTACTS AND LOCATIONS:
Locations (1):
- MTI-Mardan Medical Complex, Mardan, Khyber Pakhtunkhwa, Pakistan